CLINICAL TRIAL: NCT05947825
Title: The Safety and Tolerance of Sitagliptin Combined With Gemcitabine and Albumin-bound Paclitaxel in Subjects With Locally Advanced and Metastatic Pancreatic Adenocarcinoma: an Open, One-Armed, Single-Center, Phase Ⅱ Study.
Brief Title: Sitagliptin Combined With Gemcitabine and Albumin-bound Paclitaxel in PDAC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sitagliptin plus AG-Tianjin
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: PDAC; sitagliptin
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Combination of sitagliptin+ gemcitabine + nab-paclitaxel (Experimental): Drug: Sitagliptin Sitagliptin will be administered orally once a day at a dose of 100 mg depending on cohort assignment.
  Drug: Gemcitabine Gemcitabine will be intravenously administered on Days 1 and 8 of every 21-day cycle at a dose of 1000 mg/m2 depending on cohort assignment.
  Drug: Nab-Paclitaxel Nab-Paclitaxel will be intravenously administered on Days 1 and 8 of every 28-day cycle at a dose of 125 mg/m2 depending on cohort assignment.
  Interventions: Drug: Combination of sitagliptin+ gemcitabine + nab-paclitaxel

INTERVENTIONS:
Drug: Combination of sitagliptin+ gemcitabine + nab-paclitaxel — Drug1: Sitagliptin will be administered orally once a day at a dose of 100 mg depending on cohort assignment.
  Drug2: Gemcitabine will be intravenously administered on Days 1 and 8 of every 21-day cycle at a dose of 1000 mg/m2 depending on cohort assignment.
  Drug3: Nab-Paclitaxel will be intravenously administered on Days 1 and 8 of every 28-day cycle at a dose of 125 mg/m2 depending on cohort assignment.

SUMMARY:
The purpose of this study is to determine the safety and tolerance of sitagliptin combined with gemcitabine and albumin-bound paclitaxel in subjects with locally advanced and metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
This is a single-institution, prospective, open, one-armed phase Ⅱ clinical trial of sitagliptin combined with gemcitabine and nab-paclitaxel. This study will enroll 30 PDAC patients over 12-15 months.

ELIGIBILITY:
Inclusion Criteria:

1.≥ 18 years old at the time of informed consent 2.Ability to provide written informed consent and HIPAA authorization 3.Untreated locally advanced or metastatic Pancreatic Ductal Adenocarcinoma (PDAC) as defined by National Comprehensive Cancer Network (NCCN) guidelines or, untreated metastatic PDAC (prior adjuvant therapy is permitted if it's been greater than 6 months since completion) 4.Histologically or cytologically confirmed PDAC 5.Confirmed PDAC that is measurable or evaluable per RECIST 1.1 6.Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 7.Gastrointestinal symptoms (nausea, vomiting, and diarrhea) of Grade 1 or less 8.Adequate organ function as defined by:

1. Aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 3 x upper limits of normal (ULN)
2. Total bilirubin level ≤ 2 x ULN
3. Creatinine level < 1.7mg/dL For patients with a Body Mass Index (BMI) > 30 kg/m2, lean body weight should be used to calculate the glomerular filtration rate (GFR).
4. Hemoglobin (Hgb) ≥ 90 g/L, Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, Platelets ≥ 80 x 109/L, Acceptable coagulation studies as demonstrated by prothrombin time (PT) within normal limits (+/-15%) unless they are on anticoagulation therapy
5. Life expectancy estimated at ≥ 3 months

Exclusion Criteria:

1. With any cancer other than PDAC in recent 5 years;
2. With myocardial infarction;
3. Uncontrolled hypertension (systolic pressure>150mmHg or diastolic pressure>100mmHg after treatment)
4. LVEF<50%
5. History of hemorrhage or thromboembolism in the last 6 months
6. Psychiatric history
7. Pregnant or breastfeeding
8. Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
9. Autoimmune disease
10. Uncontrolled active infection
11. Other drugs that must be used during the trial may affect the metabolism of the experimental drugs (Sitagliptin, gemcitabine, nab-paclitaxel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time | from start of treatment until progression or last known follow up (i.e up to 2 years)
  Rrogression-free survival time of PDAC patients

SECONDARY OUTCOMES:
Objective Response Rate | from start of treatment until 30 days after treatment discontinuation (i.e up to 2 years) Using RECIST 1.1
  Objective Response Rate
Frequency of adverse events in the safety evaluable population | Time Frame: from start of treatment until 30 days after treatment discontinuation (i.e up to 2 years)
  Frequency of adverse events in the safety evaluable population
Median Overall Survival (mOS) of the treated population | from start of treatment until death or last known follow up (i.e up to 2 years)
  Median Overall Survival (mOS) of the treated population
Disease control rate (DCR) | 8 weeks
  Disease control rate (DCR)

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Dr., Principal Investigator — Tianjin Medical University affiliated Cancer Hospital

IPD SHARING:
Plan to Share IPD: No